CLINICAL TRIAL: NCT03406169
Title: Patterns of Erectile Recovery After Robotic-Assisted Laparoscopic Prostatectomy With and Without Penile Rehabilitation
Brief Title: Erectile Recovery After Robotic-Assisted Laparoscopic Prostatectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kuwong B Mwamukonda, Staff Urologist, Brooke Army Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: C.2017.001
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Erectile Dysfunction; Prostate Cancer
Keywords: penile rehabilitation
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms | interventions — Sildenafil Citrate; Tablets; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sildenafil 25mg Oral Tablet (Active Comparator): 25mg sildenafil citrate twice daily
  Interventions: Drug: Sildenafil 25 MG Oral Tablet
- Pentoxifylline (Active Comparator): 400mg pentoxifylline twice daily
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): placebo twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil 25 MG Oral Tablet — twice a day dosing
  Other Names: viagra
  Arms: Sildenafil 25mg Oral Tablet
Drug: Pentoxifylline — 400mg twice a day
  Other Names: trental
  Arms: Pentoxifylline
Other: Placebo — placebo twice a day
  Arms: Placebo

SUMMARY:
The study is a prospective, randomized, double-blind, placebo-controlled drug study to evaluate the pattern of erectile function recovery after robotic assisted laparoscopic prostatectomy (RALP). We hope to illustrate that early and continuous therapy with either Sildenafil citrate or pentoxyfylline after nerve sparing RALP will promote improved erectile function.

DETAILED DESCRIPTION:
Evaluation of erectile function with the International Index of Erectile Function Questionnaire (IIEF) and measurement of penile length any time between the prostate biopsy and 3 days prior to RALP will be performed.

Patients will undergo a unilateral or bilateral nerve sparing-RALP.

Patients will be randomized to receive either 25mg Viagra twice daily, 400mg pentoxifylline twice daily or placebo twice daily, starting on the first postoperative day after surgery and continuing for one year. The biostatistician generates a table of random numbers. 120 subjects anticipated to enroll at Brooke Army Medical Center will be divided into 3 groups, sildenafil, pentoxifylline or placebo. The randomization table will be given to the research pharmacist.

Patients will have their erectile function evaluated at 3 months, 6 months, 9 months, and 12 months with IIEF and sexual intercourse diary. These visits are routine for post-operative care following a RALP, however, completion of the IIEF and sexual intercourse diary are being performed for study purposes.

Patients will stop therapy at 12 months and penile length will be re-measured. Measurement of penile length will be done for study purposes at the standard 1 year post-operative follow up visit.

Patient will undergo a 6 week washout period during which neither drug will be used, then repeat analysis of erectile function with IIEF will be performed, after which they may restart standard erectile dysfunction therapy as desired. This washout period and follow up will be for study purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have had a prostate biopsy positive for prostate cancer.
2. Patient must be age 30 - 89 years.
3. Patient must be willing to sign the Institutional Review Board approved consent.
4. Patient must have had (or be about to undergo) bilateral or unilateral nerve sparing RALP.
5. Patient must have an International IIEF equal to or greater than 21.

Exclusion Criteria:

1. Patients with known unstable angina, uncontrolled hypertension, congestive heart failure, or cardiovascular accident within the preceding 2 weeks.
2. Patients being treated with nitrate therapy.
3. Patients with significant renal or hepatic impairment, cerebrovascular disease.
4. Patients with prior erectile dysfunction as indicated by the initial IIEF.
5. Patients younger than 30 years of age.
6. Patients who did/will not have a unilateral or bilateral nerve sparing radical prostatectomy.
7. Patients who have had a prior reaction to Sildenafil or pentoxifylline.
8. Patients taking any potent inhibitor of cytochrome P450 3A4 (e.g., ketoconazole, itraconazole, erythromycin, etc.).
9. Patients with a clinically significant abnormality on preoperative ECG that in the opinion of the investigator may increase the patient's cardiovascular risk in this study.
10. Patients with a history of left ventricular outflow obstruction (e.g. aortic stenosis, idiopathic hypertrophic subaortic stenosis).
11. Patients with resting hypotension (BP < 90/50 mm Hg), or resting hypertension (BP > 170/110 mm Hg).
12. Patients with retinitis pigmentosa.
13. Patients with a bleeding disorder.
14. Patients with active peptic ulceration.
15. Patients with conditions that may predispose to priapism (e.g. sickle cell anemia, multiple myeloma, or leukemia).
16. Patients who have previously experienced non-arteritic ischemic optic neuropathy (NAION).

Ages: 30 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have a prostate
Enrollment: 180 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Erectile function | 12 months post surgery
  As measured by IIEF

SECONDARY OUTCOMES:
Penile length | 12 months post surgery
  Stretched length in cm from pubis to coronal ridge

CONTACTS AND LOCATIONS:
Overall Officials: Kuwong B Mwamukonda, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States